CLINICAL TRIAL: NCT06778928
Title: Posterior Wall Sparing of Laparoscopic Cholecystectomy in Cirrhotic Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Adnan mohamed, Principal investigator, Assiut University
Other Study IDs: cholecystectomy cirrhotic
Record Dates: First submitted 2024-10-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-10

CONDITIONS: Cholecystitis in Cirrhotic Patients
MeSH Terms: interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Posterior wall sparing of laparoscopic cholecystectomy in cirrhotic patients: To assess the outcome of posterior wall sparing of laparoscopic cholecystectomy in cirrhotic patient
  Interventions: Procedure: laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: laparoscopic cholecystectomy — Posterior wall sparing of laparoscopic cholecystectomy in cirrhotic patients

SUMMARY:
To assess the outcome of posterior wall sparing of laparoscopic cholecystectomy in cirrhotic patients in Assuit university hospitals and El Rajhi hospital.

DETAILED DESCRIPTION:
Cholelithiasis is found in about one third of patients with liver cirrhosis and about twice as much as in the overall population. Predisposing factors for that include functional gallbladder alterations (reduced motility and decreased emptying), reduction in bile acidity, increased unconjugated bilirubin secretion, increased levels of estrogen, and increased intravascular haemolysis due to hypersplenism. Symptomatic biliary stones in patients with liver cirrhosis are associated with higher morbidity and mortality rates than those in patients with a non-cirrhotic liver. laparoscopic cholecystectomy is the gold standard for the treatment of most of gallbladder problems because of its several advantages over open cholecystectomy including shorter convalescence period and hospital stay. Furthermore, considering its safety, it is the gold-standard procedure in selected patients with symptomatic cholelithiasis and hepatic cirrhosis, especially Child-Pugh score A and B patients. Separation of posterior wall of the gallbladder from the liver bed in cirrhotic individuals is difficult and risky during a laparoscopic cholecystectomy surgery because of high-risk gall bladder bed due to fibrosis and tortuous, dilated vessels there so the strategy is leaving the posterior wall intact with the liver and the remnant mucosa was removed either by mucosectomy in patients with acute cholecystitis or by electro fulguration in those with chronic cholecystitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 - 60 years old Child A and B cirrhotic patients with Cholelithiasis Patient fit for surgery

Exclusion Criteria:

* Patient with pervious abdominal surgery

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 60 cirrhotic patients age from 18 to 60 years who were admitted for cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Intra and Post-operative haemorrhage | Surgery then 2 days follow up
Postoperative bile leak | Surgery then 1 week follow up
Changes of liver function tests | Surgery then 1 week follow up
  AST, ALT, Billirubin
Worsening of ascites | Surgery then 1 week follow up
Port site infection | Surgery then 1 week folow up

SECONDARY OUTCOMES:
Operative time | From the end of induction of anasthesia to the closure of port site incisions
Postoperative hospital stay | surgery then up to 1 week hospital stay before discharge

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shaikh AR, Muneer A. Laparoscopic cholecystectomy in cirrhotic patients. JSLS. 2009 Oct-Dec;13(4):592-6. doi: 10.4293/108680809X12589999537959. PMID 20202403
- [Background] Schiff J, Misra M, Rendon G, Rothschild J, Schwaitzberg S. Laparoscopic cholecystectomy in cirrhotic patients. Surg Endosc. 2005 Sep;19(9):1278-81. doi: 10.1007/s00464-004-8823-z. Epub 2005 Jul 21. PMID 16021366
- [Background] Palanivelu C, Rajan PS, Jani K, Shetty AR, Sendhilkumar K, Senthilnathan P, Parthasarthi R. Laparoscopic cholecystectomy in cirrhotic patients: the role of subtotal cholecystectomy and its variants. J Am Coll Surg. 2006 Aug;203(2):145-51. doi: 10.1016/j.jamcollsurg.2006.04.019. Epub 2006 Jun 22. PMID 16864026
- [Background] Cassinotti E, Baldari L, Boni L, Uranues S, Fingerhut A. Laparoscopic Cholecystectomy in the Cirrhotic: Review of Literature on Indications and Technique. Chirurgia (Bucur). 2020 Mar-Apr;115(2):208-212. doi: 10.21614/chirurgia.115.2.208. PMID 32369724